CLINICAL TRIAL: NCT02176278
Title: Using a Diabetic Kidney Disease (DKD) Registry to Treat to Multiple Targets (TMT) (DKD-TMT)
Brief Title: Using a Diabetic Kidney Disease (DKD) Registry to Treat to Multiple Targets (TMT)
Acronym: DKD-TMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2013.609-T
Record Dates: First submitted 2014-04-28; First posted 2014-06-27 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Diabetes; Asian; Joint Asia Diabetes Evaluation (JADE) Program
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care Group (No Intervention): Usual care (UC) group:
  After undergoing a comprehensive assessment, all patients will receive UC in accordance to the practice of the health institution and return at 12 months for a repeat comprehensive assessment.
- Empowered Care Group (Experimental): Empowered care (EC) group:
  After undergoing a comprehensive assessment, all patients will be given a JADE comprehensive assessment report which is a personalize risk report with treatment targets and decision support with explanation from the doctor and nurse. In addition to receiving UC in accordance to the practice of the health institution, the nurse will provide telephone reminder to patient 3-monthly to remind them to adhere to treatment, provide support and empower them to discuss with their doctors about their treatment needs and any concerns. All patients will return at 12 month for a repeat comprehensive assessment.
  Interventions: Other: Telephone Reminder; Other: Personalized Risk Report for Patient Empowerment
- Team-based, Empowered Care Group (Experimental): Team-based, empowered care (TEC) group:
  After undergoing a comprehensive assessment, patients randomized to the TEC group will be given a JADE comprehensive assessment report which is a personalized risk report for patient empowerment. They will receive telephone reminders and doctor-nurse follow up at least 3 monthly to achieve multiple targets recommended. The patients will also be given JADE reports 3-monthly and return at 12 month for a repeat comprehensive assessment.
  Interventions: Other: Telephone Reminder; Other: Doctor-Nurse Follow Up; Other: Personalized Risk Report for Patient Empowerment

INTERVENTIONS:
Other: Telephone Reminder — Nurse will provide telephone contact to patients every 3 month to remind them to adhere to treatment, provide support and empower them to discuss with their doctors about their treatment needs and any concerns
  Arms: Empowered Care Group; Team-based, Empowered Care Group
Other: Doctor-Nurse Follow Up — Patient will be followed by a doctor-nurse team at least 3 monthly to achieve multiple targets recommended as A1c<7%, BP<130/80 mmHg, LDL-C<1.8 mmol/l, triglyceride<1.7 mmol/l and persistence with RAS inhibitors taking into consideration safety and tolerability (e.g. hypoglycemia, hypotension, changes in electrolytes). Patient report will be given after follow up.
  Arms: Team-based, Empowered Care Group
Other: Personalized Risk Report for Patient Empowerment — Patients will be given with personalized risk reports after baseline and 12-month repeat comprehensive assessments.
  Arms: Empowered Care Group; Team-based, Empowered Care Group

SUMMARY:
In this quality improvement program (DKD-TMT), patients will be recruited from multiple sites across Asia, with each site recruiting at least 300 type 2 diabetic patients with Diabetic Kidney Disease (DKD). After explanation by trained doctors and nurses, and with written informed consent, patients will be randomized to the UC (n=100, usual care) group, the EC (n=100, empowered care) group, or the TEC (n=100, team-based, empowered care) group. Patients in all 3 groups will undergo a comprehensive assessment (CA) guided by the templates in the Joint Asia Diabetes Evaluation (JADE) portal at baseline and at month 12. They will also self-administer a set of questionnaires for assessing quality of life and psychological distress during the CA at both time points.

During the 12 months between the 2 CAs:

* Patients in the UC group will receive UC in accordance to the practice of the health institution.
* Patients in the EC group will receive a JADE summary report with personalized risk prediction, treatment targets and decision support with explanation from the doctor and nurse. In addition to receiving UC in accordance to the practice of the health institution, the nurse will telephone the patient 3-monthly to remind them to adhere to treatment, provide support and empower them to discuss with their doctors about their treatment needs and any concerns.
* Patients in the TEC group will be followed by a doctor-nurse team at least 3 monthly to achieve multiple targets, but tailored to patients' risk profile. The patients will receive telephone reminders and also be given a JADE follow up report 3-monthly.

The primary composite endpoint is attainment of treatment goals and/or control of risk factors. The secondary composite endpoint is all-diabetes related clinical endpoints. The tertiary changes are behavioral changes, psychological well-being and quality of life.

DETAILED DESCRIPTION:
Hypothesis: Patient empowerment and team-based care augmented by the JADE program with features of risk stratification and decision support improves multiple risk factor control in Asian type 2 diabetic patients with chronic kidney disease. Attaining multiple treatment targets reduces all diabetes-related endpoints in these high risk patients.

Objectives: To use the JADE program which 1) includes task delegation and change in workflow augmented by 2) a web-based portal consisting of features of risk stratification, feedback, recommendations and decision support to set up a DKD registry in order to 1) document control of risk factors and care standards in real practice in Asian type 2 diabetic patients; 2) empower doctors and patients to make informed decisions and 3) use a team approach to treat to multiple targets and reduce all diabetes related clinical outcomes.

Study design: This will be a multicentre randomized translational program to compare the effects of usual care (UC) versus empowered care (EC) versus team-based, empowered care (TEC) on risk factor control and clinical outcomes in 3000 patients with DKD in Asian countries.

Intervention: All patients will undergo a comprehensive assessment (CA) guided by the templates in the JADE portal at baseline and at month 12. All patients will also self-administer a set of questionnaires for assessing quality of life (EQ-5D-3L, WHOQOL-BREF, and a Time Trade-Off (TTO) question) and psychological distress (PHQ-9 and DASS-21) during the CA at baseline and at month 12.

During the 12 months between the 2 CAs:

* Patients in the UC group will receive UC in accordance to the practice of the health institution.
* Patients in the EC group will receive a JADE summary report with personalized risk prediction, treatment targets and decision support with explanation from the doctor and nurse. In addition to receiving UC in accordance to the practice of the health institution, the nurse will telephone the patient 3-monthly to remind them to adhere to treatment, provide support and empower them to discuss with their doctors about their treatment needs and any concerns.
* Patients in the TEC group will be followed by a doctor-nurse team at least 3 monthly to achieve multiple targets, but tailored to patients' risk profile. The patients will receive telephone reminders and also be given a JADE follow up report 3-monthly.

Outcome: The primary composite endpoint is attainment of treatment goals and/or control of risk factors. The secondary composite endpoint is all-diabetes related clinical endpoints. The tertiary changes are behavioral changes, psychological well-being and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with serum creatinine above 30% upper limit of normal of the laboratory range and/or estimated glomerular filtration rate (eGFR)< 65ml/min/1.73m2; or type 2 diabetic patients with both eGFR between 60 to 90ml/min/1.73m2 and urine albumin creatinine ratio (ACR) ≥ 25 mg/mmol.
* Willingness to return for regular follow up visits

Exclusion Criteria:

* Inability to give informed consent
* Life threatening condition with reduced life expectancy
* Patients on dialysis or eGFR<15 ml/min/1.732

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Attainment of at least 3 treatment targets | 1 year
  Attainment of at least 3 treatment targets of
  * A1c<7%
  * BP<130/80 mmHg
  * LDL-C<1.8 mmol/L
  * Triglyceride<1.7 mmol/L
  * Persistence with RAS inhibitors taking into consideration safety and tolerability (e.g. hypoglycemia, hypotension, changes in electrolytes)

SECONDARY OUTCOMES:
Incidence of all-diabetes related endpoints | 1 year
  Incidence of all-diabetes related endpoints (vascular, cancer, non-vascular non-cancer and all-cause death) between patients who attain at least 3 targets versus those who do not

OTHER OUTCOMES:
Changes in A1c | 1 Year
  To examine the absolute and % changes in A1c amongst the UC, EC and TEC groups
Changes in eGFR | 1 Year
  To examine the absolute and % changes in eGFR amongst the UC, EC and TEC groups
Use of medication | 1 year
  To understand the use of medications including statins, RAS inhibitors and insulin amongst the UC, EC and TEC groups
Incidence of ESRD and all-cause death | 1 year
  To examine the difference of incidence of ESRD and all-cause death between patients who are treated to multiple targets and those who are not
Incidence of all CV events | 1 year
  To investiage the difference of incidence of all CV events including stroke, acute myocardial infarction, heart failure, acute coronary syndrome, all-cause death between patients who are treated to multiple targets and those who are not
Incidence of all-site cancer and all-cause death | 1 year
  To examine incidence of all-site cancer and all-cause death between patients who are treated to multiple targets and those who are not
Cost-effectiveness and quality of life analysis | 1 year
Changes in lipid | 1 year
  To examine the absolute and % changes in lipids amongst the UC, EC and TEC groups
Changes in BP | 1 year
  To examine the absolute and % changes in BP amongst the UC, EC and TEC groups
Changes in body weight | 1 year
  To exmine the absolute and % changes in body weight amongst the UC, EC and TEC groups
Changes in albuminuria | 1 year
  To exmine the absolute and % changes albuminuria amongst the UC, EC and TEC groups

CONTACTS AND LOCATIONS:
Overall Officials: Juliana CN Chan, MD, Principal Investigator — Asia Diabetes Foundation
Locations (11):
- The Forth Affiliated Hospital of China Medical University, Shengyang, China
- Hong Kong (2):
  - Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - Department of Medicine, Alice Ho Miu Ling Nethersole Hospital, Hong Kong
- Malaysia (2):
  - Universiti Sains Malysia, Kubang Kerian, Kelantan
  - University Malaya Medical Centre, University of Malaya, Kuala Lumpur
- South Korea (3):
  - Bucheon St. Mary's Hospital, The Catholic University of Korea, Seoul, Gyenonggo-do
  - Hally University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Seoul St.Mary's Hospital, The Catholic Unviersity of Korea, Seoul
- Taipei Veterans General Hospital, Taipei, Taiwan
- Theptarin Hospital, Bangkok, Thailand
- Hoa Hao MEDIC Company LMT, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan J, So W, Ko G, Tong P, Yang X, Ma R, Kong A, Wong R, Le Coguiec F, Tamesis B, Wolthers T, Lyubomirsky G, Chow P. The Joint Asia Diabetes Evaluation (JADE) Program: a web-based program to translate evidence to clinical practice in Type 2 diabetes. Diabet Med. 2009 Jul;26(7):693-9. doi: 10.1111/j.1464-5491.2009.02751.x. PMID 19573118
- [Background] Chan JC, So WY, Yeung CY, Ko GT, Lau IT, Tsang MW, Lau KP, Siu SC, Li JK, Yeung VT, Leung WY, Tong PC; SURE Study Group. Effects of structured versus usual care on renal endpoint in type 2 diabetes: the SURE study: a randomized multicenter translational study. Diabetes Care. 2009 Jun;32(6):977-82. doi: 10.2337/dc08-1908. PMID 19460913
- [Background] Wu JY, Leung WY, Chang S, Lee B, Zee B, Tong PC, Chan JC. Effectiveness of telephone counselling by a pharmacist in reducing mortality in patients receiving polypharmacy: randomised controlled trial. BMJ. 2006 Sep 9;333(7567):522. doi: 10.1136/bmj.38905.447118.2F. Epub 2006 Aug 17. PMID 16916809
- [Background] Leung WY, So WY, Tong PC, Chan NN, Chan JC. Effects of structured care by a pharmacist-diabetes specialist team in patients with type 2 diabetic nephropathy. Am J Med. 2005 Dec;118(12):1414. doi: 10.1016/j.amjmed.2005.07.050. PMID 16378791
- [Background] Leung WY, So WY, Tong PC, Lo MK, Lee KF, Ko GT, Chan WB, Cockram CS, Brenner BM, Shahinfar S, Critchley JA, Chan JC. The renoprotective effects of structured care in a clinical trial setting in type 2 diabetic patients with nephropathy. Nephrol Dial Transplant. 2004 Oct;19(10):2519-25. doi: 10.1093/ndt/gfh408. Epub 2004 Jul 27. PMID 15280527
- [Background] Chan JC, Sui Y, Oldenburg B, Zhang Y, Chung HH, Goggins W, Au S, Brown N, Ozaki R, Wong RY, Ko GT, Fisher E; JADE and PEARL Project Team. Effects of telephone-based peer support in patients with type 2 diabetes mellitus receiving integrated care: a randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):972-81. doi: 10.1001/jamainternmed.2014.655. PMID 24781960
- [Derived] Chan JCN, Thewjitcharoen Y, Nguyen TK, Tan A, Chia YC, Hwu CM, Jian D, Himathongkam T, Wong KL, Choi YM, Mirasol R, Mohamed M, Kong APS, Ma RCW, Chow EYK, Ozaki R, Lau V, Fu AWC, Hong EG, Yoon KH, Tsang CC, Lau ESH, Lim LL, Luk AOY. Effect of a Web-Based Management Guide on Risk Factors in Patients With Type 2 Diabetes and Diabetic Kidney Disease: A JADE Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e223862. doi: 10.1001/jamanetworkopen.2022.3862. PMID 35333363
- See also: Asia Diabetes Foundation — https://www.adf.org.hk